CLINICAL TRIAL: NCT05277168
Title: AN OPEN-LABEL, SINGLE-ARM, MULTI-CENTER PHASE I/IIA CLINICAL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF SHR-A1904 IN SUBJECTS WITH ADVANCED SOLID TUMORS
Brief Title: A TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF SHR-A1904 IN SUBJECTS WITH ADVANCED SOLID TUMORS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1904-I-104
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: SHR-A1904 in Subjects with Advanced Solid tumors
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm : SHR-A1904
  Interventions: Drug: SHR-A1904

INTERVENTIONS:
Drug: SHR-A1904 — Single Arm ：It is a dose-escalation and dose-expansion study of SHR-A1904 in subjects with advanced solid tumors

SUMMARY:
The study (dose escalation/expansion) is being conducted to assess the safety and tolerability of SHR-A1904 in subjects with advanced solid tumors, and to determine maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D), to assess preliminary efficacy of SHR-A1904, pharmacokinetic (PK) profile and immunogenicity of SHR-A1904 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated ICF indicating that the subject has been informed of all pertinent aspects of the study.
2. Age >18.
3. ECOG performance status of 0-1.
4. Life expectancy of ≥3 months.
5. Subjects with pathologically diagnosed advanced relapsed or refractory solid tumors, either gastric and gastroesophageal junction (GEJ) cancer, or pancreatic cancer, who are intolerable to SoC, have progressed through all available treatment options, or for whom there is no efficacious treatment available. Subjects must have pathological classification (e.g., adenocarcinoma etc.) documented.
6. Positive expression of Claudin 18.2 (>=50% of cells with 2+ or 3+ expression, either from fresh or archival tissue) is required prior to enrollment and participation in this study. Positivity for Claudin 18.2 is defined as tumor cells showing partial or complete membrane staining. The percentage of tumor cells at four different staining intensities will be estimated: 0 (no staining), 1+ (weak), 2+ (moderate), and 3+ (strong). The sum of all 4 percentages should equal 100%. The H-score is determined according to the H-Score formula: [1 x Percentage of tumor cells stained at 1+] + [2 x Percentage of tumor cells stained at 2+] + [3 x Percentage of tumor cells stained at 3+] = H-Score (range 0 or 1-300). Actual figure of Claudin 18.2 expression tested by IHC should be documented. Subjects must have pathological classification (e.g., adenocarcinoma) documented.
7. Has at least one measurable lesion as defined by RECIST v1.1.
8. Has adequate organ and bone marrow function within 7 days prior to administration of study treatment defined below: with no blood transfusion or hematopoietic growth factor support within 2 weeks prior to screening): • Absolute neutrophil count (ANC) ≥1.5 × 109 /L • Platelet count (PLT) ≥100 × 109 /L • Hemoglobin (Hb) ≥90 g/L • TBIL ≤1.5 × ULN • ALT and AST ≤3 × ULN (≤5 × ULN for liver metastasis) • Creatinine clearance ≥60 mL/min/1.73 m2 based on Cockcroft-Gault equation (Appendix 5) • Activated partial thromboplastin time (APTT) and prothrombin time (PT) ≤1.5 × ULN. • Fridericia-corrected QT interval (QTcF) ≤450 msec. If ECG demonstrates QTc >450 msec at screening, an ECG re-examination is allowed, and subjects will be eligible if it demonstrates QTc ≤ 450 msec. • LVEF ≥50%.
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 3 days before the first dose. WOCBP and male subjects whose partners are WOCBP must agree to use effective contraception method during the study period and within 5 half-lives of SHR-A1904 + 6 months after the last dose of SHR-A1904. (see Appendix 2 for details).

Exclusion Criteria:

1. Plan to receive any other anti-tumor treatments during the treatment period of this study.
2. Subjects participated in a prior investigational study or received anticancer treatment, and have not recovered from side effects of such therapy.
3. Underwent major surgical operation within 4 weeks before the first dose of this IP.
4. Received treatments with strong CYP3A4, CYP2D6, P-gp, or BCRP inhibitors or inducers within < 5 half-lives of the drug before the first dose of the study.
5. Previously received total gastrectomy (only for subjects of the dose-escalation part.
6. Adverse events caused by previous anti-tumor treatments have not recovered to Grade ≤1 according to NCI-CTCAE 5.0 (except for alopecia; some tolerable chronic Grade 2 toxicities may also be excluded as judged by the investigator after consultation with the sponsor).
7. Known to be allergic to any component of SHR-A1904 product (antibody conjugated toxin, antibody), or allergic to humanized monoclonal antibody products.
8. Subjects with known brain metastases, unless the participant is > 1 month from definitive therapy (surgery or radiotherapy), has no evidence of tumor growth on an imaging study and is clinically stable with respect to the tumor at the start of study intervention.
9. Subjects with a second primary cancer, except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, and other solid tumors curatively treated with no evidence of disease for ≥3 years prior to the first dose of the study.
10. Class III-IV cardiac insufficiency as per the New York Heart Association (NYHA) criteria; arrhythmia requiring long-term drug control; unstable angina or acute myocardial infarction within 6 months before the first dose of the study.
11. Subjects with a history of clinically significant lung diseases (e.g., interstitial pneumonia, radiation pneumonia, and pulmonary fibrosis) or who are suspected to have these diseases by chest imaging at screening period.
12. Serious infections that require use of intravenous antibiotics, antiviral drugs, or antifungal drugs during the study period.
13. Hepatitis B (HBV, chronic or acute; defined as having a known positive hepatitis B surface antigen [HbsAg] test at the time of screening) or hepatitis C (HCV) infection requiring treatment
14. Has a history of immunodeficiency (including positive results of HIV test in screening, and other acquired and congenital immunodeficiencies) or organ transplant.
15. Presence of accompanying diseases (such as poorly controlled hypertension, serious diabetes mellitus, thyroid disorder, psychosis, etc.) that may pose serious risks to the safety of the subject or may affect the subject's ability to complete the study, or any other situation as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | the first cycle of administration, up to 21 days
  DLT is defined during the first cycle of the study treatment and assessed as certainly or at least possibly related to SHR-A1904 treatment.
Maximum tolerated dose (MTD) | the first cycle of administration, up to 21 days
  defined as the dose with the estimated toxicity probability which is the closest to the target toxicity probability.
Recommended Phase 2 Dose (RP2D) | the first cycle of administration, up to 21 days
  RP2D is the dose selected for further study based on the phase I study results.
Adverse events (AEs) and serious adverse events (SAEs) | from the signing of informed consent form to the end of safety follow-up period (90 days after the last dose)

SECONDARY OUTCOMES:
Objective response rate (ORR) | evaluated until the end of study, approximately 12 months after the first dose of study drug of the last subject, currently estimated March 2026
  The proportion of efficacy evaluable subjects with the best overall response (BOR) of CR or PR as per RECIST 1.1 criteria.
Duration of response (DoR) | evaluated until the end of study, approximately 12 months after the first dose of study drug of the last subject
  defined as the time from first documented tumor response (CR/PR) until PD/death.
Clinical benefit rate (CBR) | evaluated until the end of study, approximately 12 months after the first dose of study drug of the last subject
  defined as the percentage of subjects who have achieved complete response (CR), partial response (PR) and/or stable disease (SD) lasting over 24 weeks (CR+PR+SD≥24 weeks).
Progression-free survival (PFS) | evaluated until the end of study, approximately 12 months after the first dose of study drug of the last subject
  defined as the time from the first dose until PD/death.
Overall survival (OS) | until the end of study, approximately 12 months after the first dose of study drug of the last subject
  defined as the time from first dose of study drug until death from any cause.
Time to maximum concentration (Tmax) | up to 30 days after the last dose
Maximum concentration (Cmax) | up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (28):
- United States (7):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - LSU Health Sciences Center, New Orleans, Louisiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health, Greenville, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (9):
  - Central Coast Local Health District, Gosford, New South Wales
  - Sydney South West Private Hospital, Liverpool, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Genesis Care North Shore, St Leonards, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gold Coast Private Hospital, Southport, Queensland
  - Peninsula and South Eastern Haematology & Oncology Group (PASO), Frankston, Victoria
  - One Clinical Research (OCR), Nedlands, Western Australia
- National Institute of Oncology, Arensia Research Clinic, Chisinau, Moldova
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam
  - CHA Bundang Medical Centre, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided